CLINICAL TRIAL: NCT01352845
Title: A Phase 3, Randomized, Placebo-controlled, Observer-blinded, Trial To Assess The Safety, Tolerability, And Immunogenicity Of Bivalent Rlp2086 Vaccine When Administered As A 3-dose Regimen In Healthy Young Adults Aged >=18 To <26 Years
Brief Title: A Trial to Assess the Safety, Tolerability, and Immunogenicity of Bivalent rLP2086 Vaccine When Given to Healthy Young Adults Aged >=18 to <26 Years.
Acronym: B1971016
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1971016; 6108A1-2004 (Other: Alias Study Number); 2009-014492-46 (EudraCT Number)
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — factor H-binding protein, Neisseria meningitidis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rLP2086 (Experimental)
  Interventions: Biological: rLP2086
- Control (Placebo Comparator): Steril normal saline solution
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: rLP2086 — 0.5 mL dose, given at 0, 2 and 6 months
  Arms: rLP2086
Other: Placebo — 0.5 mL dose, given at 0, 2 and 6 months
  Arms: Control

SUMMARY:
This study is looking at a new vaccine that might prevent meningococcal disease, and will study the immune response elicited by this vaccine when given to healthy young adults. The study will also look at the safety of the new vaccine as well as how it is tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged >=18 and <26 years at the time of enrollment.
2. Healthy subject as determined by medical history, physical examination, and judgment of the investigator.
3. Negative urine pregnancy test for all female subjects.

Exclusion Criteria:

1. Previous vaccination with any meningococcal serogroup B vaccine.
2. Subjects who are scheduled to receive 1 or more doses of an HPV vaccine as part of a 3-dose series during the period between Visit 1 and 28 days after the second vaccination.
3. Subjects receiving any allergen immunotherapy with a nonlicensed product or receiving allergen immunotherapy with a licensed product and are not on stable maintenance doses.
4. A known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired defects in B cell function, those receiving chronic systemic (oral, intravenous, or intramuscular) corticosteroid therapy, or those receiving immunosuppressive therapy. Subjects in the United States with terminal complement deficiency are excluded from participation in this study.
5. Significant neurological disorder or history of seizure (excluding simple febrile seizure).
6. Current chronic use of systemic antibiotics.
7. Received any investigational vaccines, drugs, or devices within 28 days before administration of the first study vaccination.
8. Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3301 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (34):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Clinical Research Advantage, Inc./Desert Clinical Research, LLC, Mesa, Arizona
  - Clinical Research Advantage, Inc./ Fiel Family and Sports Medicine, PC, Tempe, Arizona
  - Anaheim Clinical Trials LLC, Anaheim, California
  - eStudySite, La Mesa, California
  - Benchmark Research, Sacramento, California
  - Broward Research Group, Hollyood, Florida
  - Altus Research Inc., Lake Worth, Florida
  - Miami Research Associates, South Miami, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Johnson County Clin-Trials, Inc., Lenexa, Kansas
  - Benchmark Research, Metairie, Louisiana
  - Milford Emergency Associates, Inc., Milford, Massachusetts
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Bellevue Urgent Care, Bellevue, Nebraska
  - Meridian Clinical Research, Bellevue, Nebraska
  - Pioneer Clinical Research, LLC, Bellevue, Nebraska
  - Meridian Clinical Research,, Omaha, Nebraska
  - Central New York Clinical Research, Manlius, New York
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Community Research, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - PEAK Research, LLC, Upper Saint Clair, Pennsylvania
  - Coastal Medical, East Greenwich, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Research Across America, Dallas, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Research Across America, Katy, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Premier Clinical Research, Spokane, Washington
- Canada (9):
  - Dr. Calvin Powell Professional Medical Corporation, Bay Roberts, Newfoundland and Labrador
  - Canadian Center for Vaccinology - IWK Health Centre, Halifax, Nova Scotia
  - Milestone Research, London, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Devonshire Clinical Research Inc., Woodstock, Ontario
  - McGill University Health Centre - Vaccine Study Centre, Pierrefonds, Quebec
  - Centre hospitalier universitaire de Québec, Québec, Quebec
  - Pro-Recherche Inc., Saint Romuald, Quebec
  - Clinique Medicale St-Louis Inc., Sainte-Foy, Québec, Quebec
- Aarhus Universitetshospital Skejby, Aarhus N, Denmark
- Finland (4):
  - Espoo Vaccine Research Clinic, Espoo
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Kokkola Vaccine Research Clinic, Kokkola
  - Seinäjoki Vaccine Research Clinic, Seinäjoki
- Poland (3):
  - NZOZ Centrum Medyczne Graniczna Sp. z o.o., Katowice
  - Specjalistyczna Poradnia Medyczna Przyladek Zdrowia, Krakow
  - NZOZ Salmed s.c., Łęczna
- Spain (6):
  - CAP Balenya, Balenya, Barcelona
  - CAP Centelles, Centelles, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - CAP El Remei, Vic, Barcelona
  - FOM (Fundacion Oftalmologica del Mediterraneo) - FISABIO, Valencia, Valencia
  - Hospital Clinic de Barcelona, Barcelona

REFERENCES:
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991
- [Derived] Beeslaar J, Absalon J, Anderson AS, Eiden JJ, Balmer P, Harris SL, Jones TR, O'Neill RE, Pregaldien JL, Radley D, Maansson R, Ginis J, Srivastava A, Perez JL. MenB-FHbp Vaccine Protects Against Diverse Meningococcal Strains in Adolescents and Young Adults: Post Hoc Analysis of Two Phase 3 Studies. Infect Dis Ther. 2020 Sep;9(3):641-656. doi: 10.1007/s40121-020-00319-0. Epub 2020 Jul 22. PMID 32700260
- [Derived] Beeslaar J, Peyrani P, Absalon J, Maguire J, Eiden J, Balmer P, Maansson R, Perez JL. Sex, Age, and Race Effects on Immunogenicity of MenB-FHbp, A Bivalent Meningococcal B Vaccine: Pooled Evaluation of Clinical Trial Data. Infect Dis Ther. 2020 Sep;9(3):625-639. doi: 10.1007/s40121-020-00322-5. Epub 2020 Jul 17. PMID 32681472
- [Derived] Ostergaard L, Vesikari T, Absalon J, Beeslaar J, Ward BJ, Senders S, Eiden JJ, Jansen KU, Anderson AS, York LJ, Jones TR, Harris SL, O'Neill R, Radley D, Maansson R, Pregaldien JL, Ginis J, Staerke NB, Perez JL; B1971009 and B1971016 Trial Investigators. A Bivalent Meningococcal B Vaccine in Adolescents and Young Adults. N Engl J Med. 2017 Dec 14;377(24):2349-2362. doi: 10.1056/NEJMoa1614474. PMID 29236639
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1971016&StudyName=A%20Trial%20to%20Assess%20the%20Safety%2C%20Tolerability%2C%20and%20Immunogenicity%20of%20Bivalent%20rLP2086%20Vaccine%20When%20Given%20to%20Healthy%20Young%20Adults%20Aged%20greater%20than%3D18%20to%20less%20than26%20Years

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 3304 participants were randomized in this study, out of which 3293 participants received vaccination.
Groups:
- Group 1 rLP2086: Recombinant lipoprotein 2086 (rLP2086) vaccine on a 0-, 2-, 6- month schedule.
- Group 2 Saline: Saline on a 0-, 2-, 6- month schedule.
Period: Overall Study
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Started | 2471 | 822
Completed | 1800 | 619
Not Completed | 671 | 203
Not completed — Lost to Follow-up | 313 | 92
Not completed — No Longer Willing to Participate | 205 | 58
Not completed — Withdrawal by Subject | 48 | 16
Not completed — No Longer Meets Eligibility Criteria | 24 | 11
Not completed — Pregnancy | 27 | 7
Not completed — Adverse Event | 22 | 6
Not completed — Other | 17 | 7
Not completed — Protocol Violation | 12 | 6
Not completed — Death | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all the participants who received at least 1 dose of the investigational product (rLP2086 or saline) and had safety data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 rLP2086 | Group 2 Saline | Total
Number analyzed (Participants) | 2471 | 822 | 3293
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.47 (2.14) | 21.52 (2.20) | 21.48 (2.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1452 | 482 | 1934
  Male | 1019 | 340 | 1359

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Greater Than or Equal to(>=)4 Fold Rise in Serum Bactericidal Assay Using Human Complement(hSBA) for 4 Primary Strains and Composite Response (hSBA>=Lower Limit of Quantification for All 4 Primary Strains Combined):Group 1
Description: Here, N signifies participants with valid and determinate hSBA titers for given strain at specified time point. This outcome measure was planned to be analyzed for Group 1 only.
Time Frame: One month after third bivalent rLP2086 vaccination
Population: Evaluable immunogenicity population: all eligible participants randomized, who received correct investigational product, had pre/post vaccination blood drawn at pre-specified time points, had valid and determinate assay results for proposed analysis, received no prohibited treatment or prohibited vaccines, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 1723
Percentage of participants
  Composite hSBA response (N=1664) | 84.9 [83.1 to 86.6]
  PMB80 [A22] (N=1695) | 80.5 [78.6 to 82.4]
  PMB2001 [A56] (N=1642) | 90.0 [88.4 to 91.4]
  PMB2948 [B24] (N=1675) | 79.3 [77.3 to 81.2]
  PMB2707 [B44] (N=1696) | 79.6 [77.6 to 81.5]

2. Primary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions (LRs) Within 7 Days After First Vaccination
Time Frame: Within 7 days after first vaccination
Population: Safety population for first vaccination included all participants who received the first dose of investigational product (rLP2086 or saline) and for whom safety information was available from first vaccination until prior to second vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2425 | 798
Percentage of participants
  Pain at injection site: Any | 84.2 [82.7 to 85.6] | 11.8 [9.6 to 14.2]
  Pain at injection site: Mild | 42.3 [40.3 to 44.3] | 10.7 [8.6 to 13.0]
  Pain at injection site: Moderate | 37.1 [35.1 to 39.0] | 1.1 [0.5 to 2.1]
  Pain at injection site: Severe | 4.8 [4.0 to 5.8] | 0.0 [0.0 to 0.5]
  Redness: Any | 13.8 [12.5 to 15.3] | 0.6 [0.2 to 1.5]
  Redness: Mild | 5.8 [4.9 to 6.8] | 0.5 [0.1 to 1.3]
  Redness: Moderate | 7.1 [6.1 to 8.2] | 0.0 [0.0 to 0.5]
  Redness: Severe | 0.9 [0.6 to 1.4] | 0.1 [0.0 to 0.7]
  Swelling: Any | 15.5 [14.1 to 17.1] | 0.6 [0.2 to 1.5]
  Swelling: Mild | 8.5 [7.4 to 9.7] | 0.3 [0.0 to 0.9]
  Swelling: Moderate | 6.8 [5.8 to 7.9] | 0.3 [0.0 to 0.9]
  Swelling: Severe | 0.2 [0.1 to 0.5] | 0.1 [0.0 to 0.7]

3. Primary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions (LRs) Within 7 Days After Second Vaccination
Time Frame: Within 7 days after second vaccination
Population: Safety population for second vaccination included all participants who received the second dose of investigational product (rLP2086 or saline) and for whom safety information was available from second vaccination until prior to third vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2076 | 706
Percentage of participants
  Pain at injection site: Any | 79.3 [77.5 to 81.1] | 7.8 [5.9 to 10.0]
  Pain at injection site: Mild | 42.2 [40.1 to 44.4] | 6.8 [5.1 to 8.9]
  Pain at injection site: Moderate | 32.7 [30.7 to 34.8] | 1.0 [0.4 to 2.0]
  Pain at injection site: Severe | 4.4 [3.6 to 5.4] | 0.0 [0.0 to 0.5]
  Redness: Any | 11.8 [10.4 to 13.3] | 0.3 [0.0 to 1.0]
  Redness: Mild | 4.6 [3.7 to 5.6] | 0.1 [0.0 to 0.8]
  Redness: Moderate | 6.3 [5.3 to 7.4] | 0.0 [0.0 to 0.5]
  Redness: Severe | 0.9 [0.6 to 1.4] | 0.1 [0.0 to 0.8]
  Swelling: Any | 14.0 [12.6 to 15.6] | 0.4 [0.1 to 1.2]
  Swelling: Mild | 7.7 [6.6 to 8.9] | 0.3 [0.0 to 1.0]
  Swelling: Moderate | 6.0 [5.0 to 7.1] | 0.1 [0.0 to 0.8]
  Swelling: Severe | 0.3 [0.1 to 0.7] | 0.0 [0.0 to 0.5]

4. Primary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions (LRs) Within 7 Days After Third Vaccination
Time Frame: Within 7 days after third vaccination
Population: Safety population for third vaccination included all participants who received the third dose of investigational product (rLP2086 or saline) and for whom safety information was available from third vaccination until post third-vaccination blood draw.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 1823 | 624
Percentage of participants
  Pain at injection site: Any | 80.4 [78.5 to 82.2] | 6.7 [4.9 to 9.0]
  Pain at injection site: Mild | 36.1 [33.9 to 38.4] | 6.4 [4.6 to 8.6]
  Pain at injection site: Moderate | 38.9 [36.6 to 41.2] | 0.3 [0.0 to 1.2]
  Pain at injection site: Severe | 5.3 [4.3 to 6.5] | 0.0 [0.0 to 0.6]
  Redness: Any | 17.1 [15.4 to 18.9] | 0.2 [0.0 to 0.9]
  Redness: Mild | 6.2 [5.1 to 7.4] | 0.2 [0.0 to 0.9]
  Redness: Moderate | 8.6 [7.3 to 9.9] | 0.0 [0.0 to 0.6]
  Redness: Severe | 2.3 [1.7 to 3.1] | 0.0 [0.0 to 0.6]
  Swelling: Any | 16.6 [14.9 to 18.4] | 0.3 [0.0 to 1.2]
  Swelling: Mild | 8.8 [7.6 to 10.2] | 0.0 [0.0 to 0.6]
  Swelling: Moderate | 7.2 [6.1 to 8.5] | 0.3 [0.0 to 1.2]
  Swelling: Severe | 0.5 [0.2 to 0.9] | 0.0 [0.0 to 0.6]

5. Primary Outcome: Percentage of Participants Reporting Systemic Events (SEs) and Antipyretic Use Within 7 Days After First Vaccination
Time Frame: Within 7 days after first vaccination
Population: Safety population for first vaccination included all participants who received the first dose of investigational product (rLP2086 or saline) and for whom safety information was available from first vaccination until prior to second vaccination. Here, 'N' signifies participants with known values reporting specific characteristic.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2425 | 798
Percentage of participants
  Fever >=38 degrees C(N=2415, 796) | 2.4 [1.8 to 3.0] | 0.6 [0.2 to 1.5]
  Fever 38 to <38.5 degreesC(N=2415, 796) | 1.6 [1.1 to 2.2] | 0.4 [0.1 to 1.1]
  Fever 38.5 to<39 degrees C(N=2415, 796) | 0.7 [0.4 to 1.2] | 0.0 [0.0 to 0.5]
  Fever 39 to 40 degrees C (N=2415, 796) | 0.0 [0.0 to 0.2] | 0.3 [0.0 to 0.9]
  Fever >40 degrees C(N=2415, 796) | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.5]
  Vomiting:Any(N=2425, 798) | 2.6 [2.0 to 3.3] | 2.1 [1.2 to 3.4]
  Vomiting:Mild(N=2425, 798) | 2.2 [1.6 to 2.8] | 2.1 [1.2 to 3.4]
  Vomiting:Moderate(N=2425, 798) | 0.4 [0.2 to 0.8] | 0.0 [0.0 to 0.5]
  Vomiting:Severe(N=2425, 798) | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.5]
  Diarrhea:Any(N=2425, 798) | 12.7 [11.4 to 14.1] | 11.8 [9.6 to 14.2]
  Diarrhea:Mild(N=2425, 798) | 10.2 [9.0 to 11.5] | 9.8 [7.8 to 12.0]
  Diarrhea:Moderate(N=2425, 798) | 2.4 [1.8 to 3.0] | 1.9 [1.1 to 3.1]
  Diarrhea:Severe(N=2425, 798) | 0.2 [0.1 to 0.5] | 0.1 [0.0 to 0.7]
  Headache:Any(N=2425, 798) | 43.9 [41.9 to 45.9] | 36.2 [32.9 to 39.7]
  Headache:Mild(N=2425, 798) | 24.3 [22.6 to 26.1] | 22.1 [19.2 to 25.1]
  Headache:Moderate(N=2425, 798) | 17.9 [16.4 to 19.5] | 13.5 [11.2 to 16.1]
  Headache:Severe(N=2425, 798) | 1.6 [1.2 to 2.2] | 0.6 [0.2 to 1.5]
  Fatigue:Any(N=2425, 798) | 50.9 [48.9 to 52.9] | 39.8 [36.4 to 43.3]
  Fatigue:Mild(N=2425, 798) | 25.4 [23.7 to 27.2] | 23.2 [20.3 to 26.3]
  Fatigue:Moderate(N=2425, 798) | 22.1 [20.5 to 23.8] | 15.8 [13.3 to 18.5]
  Fatigue:Severe(N=2425, 798) | 3.4 [2.7 to 4.2] | 0.9 [0.4 to 1.8]
  Chills:Any(N=2425, 798) | 18.1 [16.5 to 19.7] | 9.8 [7.8 to 12.0]
  Chills:Mild(N=2425, 798) | 12.0 [10.8 to 13.4] | 8.1 [6.3 to 10.3]
  Chills:Moderate(N=2425, 798) | 4.9 [4.1 to 5.8] | 1.6 [0.9 to 2.8]
  Chills: Severe(N=2425, 798) | 1.1 [0.7 to 1.6] | 0.0 [0.0 to 0.5]
  Muscle pain:Any(N=2425,798) | 25.9 [24.1 to 27.6] | 14.5 [12.2 to 17.2]
  Muscle pain:Mild(N=2425,798) | 13.0 [11.7 to 14.4] | 9.6 [7.7 to 11.9]
  Muscle pain:Moderate(N=2425,798) | 11.3 [10.0 to 12.6] | 4.4 [3.1 to 6.0]
  Muscle pain:Severe(N=2425,798) | 1.6 [1.1 to 2.2] | 0.5 [0.1 to 1.3]
  Joint pain:Any(N=2425,798) | 19.6 [18.1 to 21.3] | 10.9 [8.8 to 13.3]
  Joint pain:Mild(N=2425,798) | 10.3 [9.1 to 11.6] | 6.9 [5.2 to 8.9]
  Joint pain:Moderate(N=2425,798) | 7.9 [6.8 to 9.0] | 3.5 [2.3 to 5.0]
  Joint pain: Severe(N=2425,798) | 1.4 [1.0 to 2.0] | 0.5 [0.1 to 1.3]
  Antipyretic medication(N=2425,798) | 13.4 [12.1 to 14.8] | 8.9 [7.0 to 11.1]

6. Primary Outcome: Percentage of Participants Reporting Systemic Events (SEs) and Antipyretic Use Within 7 Days After Second Vaccination
Time Frame: Within 7 days after second vaccination
Population: Safety population for second vaccination included all participants who received the second dose of investigational product (rLP2086 or saline) and for whom safety information was available from second vaccination until prior to third vaccination. Here, 'N' signifies participants with known values reporting specific characteristic.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2076 | 706
Percentage of participants
  Fever >=38 degrees C(N=2067, 705) | 1.2 [0.7 to 1.7] | 1.0 [0.4 to 2.0]
  Fever 38 to <38.5 degreesC(N=2067, 705) | 0.7 [0.4 to 1.1] | 0.6 [0.2 to 1.4]
  Fever 38.5 to<39 degrees C(N=2067, 705) | 0.4 [0.2 to 0.8] | 0.3 [0.0 to 1.0]
  Fever 39 to 40 degrees C (N=2067, 705) | 0.1 [0.0 to 0.3] | 0.1 [0.0 to 0.8]
  Fever >40 degrees C(N=2067, 705) | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.5]
  Vomiting:Any(N=2076, 706) | 2.1 [1.5 to 2.8] | 1.6 [0.8 to 2.8]
  Vomiting:Mild(N=2076, 706) | 1.6 [1.1 to 2.3] | 1.3 [0.6 to 2.4]
  Vomiting:Moderate(N=2076, 706) | 0.5 [0.2 to 0.9] | 0.3 [0.0 to 1.0]
  Vomiting:Severe(N=2076, 706) | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.5]
  Diarrhea:Any(N=2076, 706) | 8.6 [7.4 to 9.9] | 8.1 [6.2 to 10.3]
  Diarrhea:Mild(N=2076, 706) | 6.4 [5.3 to 7.5] | 4.7 [3.2 to 6.5]
  Diarrhea:Moderate(N=2076, 706) | 1.7 [1.2 to 2.4] | 2.8 [1.7 to 4.3]
  Diarrhea:Severe(N=2076, 706) | 0.5 [0.3 to 0.9] | 0.6 [0.2 to 1.4]
  Headache:Any(N=2076, 706) | 33.1 [31.1 to 35.2] | 24.9 [21.8 to 28.3]
  Headache:Mild(N=2076, 706) | 18.4 [16.8 to 20.1] | 13.6 [11.2 to 16.3]
  Headache:Moderate(N=2076, 706) | 13.3 [11.9 to 14.8] | 10.1 [7.9 to 12.5]
  Headache:Severe(N=2076, 706) | 1.4 [1.0 to 2.1] | 1.3 [0.6 to 2.4]
  Fatigue:Any(N=2076, 706) | 39.2 [37.1 to 41.3] | 27.3 [24.1 to 30.8]
  Fatigue:Mild(N=2076, 706) | 20.6 [18.8 to 22.4] | 13.9 [11.4 to 16.7]
  Fatigue:Moderate(N=2076, 706) | 16.4 [14.8 to 18.0] | 11.5 [9.2 to 14.1]
  Fatigue:Severe(N=2076, 706) | 2.2 [1.6 to 2.9] | 2.0 [1.1 to 3.3]
  Chills:Any(N=2076, 706) | 12.4 [11.0 to 13.9] | 8.5 [6.5 to 10.8]
  Chills:Mild(N=2076, 706) | 8.1 [7.0 to 9.4] | 6.9 [5.2 to 9.1]
  Chills:Moderate(N=2076, 706) | 3.5 [2.8 to 4.4] | 1.6 [0.8 to 2.8]
  Chills: Severe(N=2076, 706) | 0.8 [0.4 to 1.2] | 0.0 [0.0 to 0.5]
  Muscle pain:Any(N=2076, 706) | 15.6 [14.0 to 17.2] | 8.5 [6.5 to 10.8]
  Muscle pain:Mild(N=2076, 706) | 7.6 [6.5 to 8.8] | 5.8 [4.2 to 7.8]
  Muscle pain:Moderate(N=2076, 706) | 7.1 [6.1 to 8.3] | 2.3 [1.3 to 3.7]
  Muscle pain:Severe(N=2076, 706) | 0.8 [0.5 to 1.3] | 0.4 [0.1 to 1.2]
  Joint pain:Any(N=2076, 706) | 15.1 [13.6 to 16.7] | 6.5 [4.8 to 8.6]
  Joint pain:Mild(N=2076, 706) | 8.1 [7.0 to 9.3] | 3.7 [2.4 to 5.3]
  Joint pain:Moderate(N=2076, 706) | 6.2 [5.2 to 7.3] | 2.5 [1.5 to 4.0]
  Joint pain: Severe(N=2076, 706) | 0.9 [0.5 to 1.4] | 0.3 [0.0 to 1.0]
  Antipyretic medication(N=2076, 706) | 12.3 [10.9 to 13.8] | 7.6 [5.8 to 9.9]

7. Primary Outcome: Percentage of Participants Reporting Systemic Events (SEs) and Antipyretic Use Within 7 Days After Third Vaccination
Time Frame: Within 7 days after third vaccination
Population: Safety population for third vaccination included all participants who received the third dose of investigational product (rLP2086 or saline) and for whom safety information was available from third vaccination until post third-vaccination blood draw. Here, 'N' signifies participants with known values reporting specific characteristic.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 1823 | 624
Percentage of participants
  Fever >=38 degrees C(N=1814, 621) | 2.0 [1.4 to 2.7] | 0.6 [0.2 to 1.6]
  Fever 38 to <38.5 degreesC(N=1814, 621) | 1.4 [0.9 to 2.0] | 0.5 [0.1 to 1.4]
  Fever 38.5 to<39 degrees C(N=1814, 621) | 0.4 [0.2 to 0.9] | 0.2 [0.0 to 0.9]
  Fever 39 to 40 degrees C (N=1814, 621) | 0.1 [0.0 to 0.4] | 0.0 [0.0 to 0.6]
  Fever >40 degrees C(N=1814, 621) | 0.1 [0.0 to 0.3] | 0.0 [0.0 to 0.6]
  Vomiting:Any(N=1823, 624) | 2.0 [1.4 to 2.7] | 1.4 [0.7 to 2.7]
  Vomiting:Mild(N=1823, 624) | 1.8 [1.2 to 2.5] | 1.1 [0.5 to 2.3]
  Vomiting:Moderate(N=1823, 624) | 0.2 [0.1 to 0.6] | 0.3 [0.0 to 1.2]
  Vomiting:Severe(N=1823, 624) | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.6]
  Diarrhea:Any(N=1823, 624) | 7.5 [6.3 to 8.8] | 6.9 [5.0 to 9.2]
  Diarrhea:Mild(N=1823, 624) | 6.1 [5.0 to 7.3] | 5.3 [3.7 to 7.3]
  Diarrhea:Moderate(N=1823, 624) | 1.2 [0.8 to 1.8] | 1.3 [0.6 to 2.5]
  Diarrhea:Severe(N=1823, 624) | 0.2 [0.0 to 0.5] | 0.3 [0.0 to 1.2]
  Headache:Any(N=1823, 624) | 32.5 [30.4 to 34.7] | 21.6 [18.5 to 25.1]
  Headache:Mild(N=1823, 624) | 17.6 [15.9 to 19.4] | 12.5 [10.0 to 15.4]
  Headache:Moderate(N=1823, 624) | 13.3 [11.8 to 15.0] | 8.3 [6.3 to 10.8]
  Headache:Severe(N=1823, 624) | 1.6 [1.1 to 2.3] | 0.8 [0.3 to 1.9]
  Fatigue:Any(N=1823, 624) | 39.3 [37.1 to 41.6] | 24.5 [21.2 to 28.1]
  Fatigue:Mild(N=1823, 624) | 18.9 [17.2 to 20.8] | 13.1 [10.6 to 16.0]
  Fatigue:Moderate(N=1823, 624) | 18.8 [17.0 to 20.6] | 9.6 [7.4 to 12.2]
  Fatigue:Severe(N=1823, 624) | 1.6 [1.1 to 2.3] | 1.8 [0.9 to 3.1]
  Chills:Any(N=1823, 624) | 12.6 [11.1 to 14.2] | 6.4 [4.6 to 8.6]
  Chills:Mild(N=1823, 624) | 7.7 [6.5 to 9.0] | 4.3 [2.9 to 6.2]
  Chills:Moderate(N=1823, 624) | 4.2 [3.3 to 5.2] | 2.1 [1.1 to 3.5]
  Chills: Severe(N=1823, 624) | 0.8 [0.4 to 1.3] | 0.0 [0.0 to 0.6]
  Muscle pain:Any(N=1823, 624) | 16.9 [15.2 to 18.7] | 7.5 [5.6 to 9.9]
  Muscle pain:Mild(N=1823, 624) | 8.9 [7.7 to 10.3] | 4.5 [3.0 to 6.4]
  Muscle pain:Moderate(N=1823, 624) | 6.8 [5.7 to 8.1] | 2.9 [1.7 to 4.5]
  Muscle pain:Severe(N=1823, 624) | 1.2 [0.7 to 1.8] | 0.2 [0.0 to 0.9]
  Joint pain:Any(N=1823, 624) | 12.6 [11.1 to 14.2] | 5.3 [3.7 to 7.3]
  Joint pain:Mild(N=1823, 624) | 6.6 [5.5 to 7.9] | 2.9 [1.7 to 4.5]
  Joint pain:Moderate(N=1823, 624) | 5.4 [4.4 to 6.5] | 2.4 [1.4 to 3.9]
  Joint pain: Severe(N=1823, 624) | 0.6 [0.3 to 1.1] | 0.0 [0.0 to 0.6]
  Antipyretic medication(N=1823, 624) | 12.8 [11.3 to 14.5] | 6.6 [4.8 to 8.8]

8. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Within 30 Days After First Vaccination
Time Frame: Within 30 days after first vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 8.62 [7.5 to 9.8] | 7.30 [5.6 to 9.3]

9. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Within 30 Days After Second Vaccination
Time Frame: Within 30 days after second vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2169 | 733
Percentage of participants | 10.10 [8.9 to 11.4] | 10.10 [8.0 to 12.5]

10. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Within 30 Days After Third Vaccination
Time Frame: Within 30 days after third vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 1889 | 649
Percentage of participants | 9.26 [8.0 to 10.7] | 7.24 [5.4 to 9.5]

11. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Within 30 Days After Any Vaccination
Time Frame: Within 30 days after any vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 21.17 [19.6 to 22.8] | 18.86 [16.2 to 21.7]

12. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) During the Vaccination Phase
Time Frame: From the first vaccination up to 1 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 31.20 [29.4 to 33.1] | 31.14 [28.0 to 34.4]

13. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After First Vaccination
Time Frame: Within 30 days after first vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 0.24 [0.1 to 0.5] | 0.12 [0.0 to 0.7]

14. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Second Vaccination
Time Frame: Within 30 days after second vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2169 | 733
Percentage of participants | 0.23 [0.1 to 0.5] | 0.00 [0.0 to 0.5]

15. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Third Vaccination
Time Frame: Within 30 days after third vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 1889 | 649
Percentage of participants | 0.11 [0.0 to 0.4] | 0.15 [0.0 to 0.9]

16. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Any Vaccination
Time Frame: Within 30 days after any vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 0.53 [0.3 to 0.9] | 0.24 [0.0 to 0.9]

17. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) During the Follow-up Phase
Time Frame: From 1 month after third vaccination up to 6 months after the third vaccination
Population: Safety population: all participants who had at least 1 dose of investigational product (rLP2086 or saline) for whom safety information was available from after post-vaccination 3 blood draw to 6 months after last study vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2067 | 704
Percentage of participants | 0.63 [0.3 to 1.1] | 0.71 [0.2 to 1.6]

18. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) During the Vaccination Phase
Time Frame: From the first vaccination up to 1 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 0.85 [0.5 to 1.3] | 0.73 [0.3 to 1.6]

19. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Throughout the Study Period
Time Frame: From the first vaccination up to 6 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 1.34 [0.9 to 1.9] | 1.34 [0.7 to 2.4]

20. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After First Vaccination
Time Frame: Within 30 days after first vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 3.89 [3.2 to 4.7] | 3.77 [2.6 to 5.3]

21. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Second Vaccination
Time Frame: Within 30 days after second vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2169 | 733
Percentage of participants | 4.66 [3.8 to 5.6] | 4.91 [3.5 to 6.7]

22. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Third Vaccination
Time Frame: Within 30 days after third vaccination
Population: Safety population for third vaccination included all participants who received the third dose of investigational product (rLP2086 or saline) and for whom safety information was available from third vaccination until until post third-vaccination blood draw.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 1889 | 649
Percentage of participants | 5.03 [4.1 to 6.1] | 3.85 [2.5 to 5.6]

23. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Any Vaccination
Time Frame: Within 30 days after any vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 10.93 [9.7 to 12.2] | 10.22 [8.2 to 12.5]

24. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE During the Vaccination Phase
Time Frame: From the first vaccination up to 1 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 19.22 [17.7 to 20.8] | 17.76 [15.2 to 20.5]

25. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE During the Follow-Up Phase
Time Frame: From 1 month after third vaccination up to 6 months after the third vaccination
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2067 | 704
Percentage of participants | 6.97 [5.9 to 8.2] | 6.68 [4.9 to 8.8]

26. Primary Outcome: Percentage of Participants Reporting at Least 1 Medically Attended Adverse Event Throughout the Study Period
Time Frame: From the first vaccination up to 6 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 21.89 [20.3 to 23.6] | 21.17 [18.4 to 24.1]

27. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After First Vaccination
Time Frame: Within 30 days after first vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 0.00 [0.0 to 0.1] | 0.00 [0.0 to 0.4]

28. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After Second Vaccination
Time Frame: Within 30 days after second vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2169 | 733
Percentage of participants | 0.23 [0.1 to 0.5] | 0.00 [0.0 to 0.5]

29. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After Third Vaccination
Time Frame: Within 30 days after third vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 1889 | 649
Percentage of participants | 0.00 [0.0 to 0.2] | 0.15 [0.0 to 0.9]

30. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After Any Vaccination
Time Frame: Within 30 days after any vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 0.20 [0.1 to 0.5] | 0.12 [0.0 to 0.7]

31. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition During the Vaccination Phase
Time Frame: From the first vaccination up to 1 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 0.32 [0.1 to 0.6] | 0.24 [0.0 to 0.9]

32. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition During the Follow-Up Phase
Time Frame: From 1 month after third vaccination up to 6 months after the third vaccination
Population: Safety population: all participants who had at least 1 dose of investigational product (rLP2086 or saline) for whom safety information was available from after post third-vaccination blood draw to 6 months after last study vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2067 | 704
Percentage of participants | 0.10 [0.0 to 0.3] | 0.00 [0.0 to 0.5]

33. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Throughout the Study Period
Time Frame: From the first vaccination up to 6 month after the third vaccination the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 0.40 [0.2 to 0.7] | 0.24 [0.0 to 0.9]

34. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate Adverse Event (AE) After First Vaccination
Time Frame: Within 30 minutes after first vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2471 | 822
Percentage of participants | 0.4 [0.2 to 0.7] | 0.6 [0.2 to 1.4]

35. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate Adverse Event (AE) After Second Vaccination
Time Frame: Within 30 minutes after second vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 2169 | 733
Percentage of participants | 0.0 [0.0 to 0.3] | 0.4 [0.1 to 1.2]

36. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate Adverse Event (AE) After Third Vaccination
Time Frame: Within 30 minutes after third vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 1889 | 649
Percentage of participants | 0.1 [0.0 to 0.3] | 0.0 [0.0 to 0.6]

37. Primary Outcome: Number of Days Participants Missed School or Work Due to AE During the Vaccination Phase
Time Frame: From the first vaccination up to 1 month after the third vaccination
Population: Safety population included all the participants who received at least 1 dose of the investigational product (rLP2086 or saline) and had safety data available. Here, number of participants analyzed signifies subjects that were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Number analyzed (Participants) | 167 | 63
Days | 5.6 (10.75) | 5.6 (13.26)

38. Secondary Outcome: Percentage of Participants With hSBA Titers >= Lower Limit of Quantification for 10 Secondary Strains Before First Vaccination and 1 Month After Third Bivalent rLP2086 Vaccination: Group 1
Time Frame: Before first vaccination, 1 month after third vaccination
Population: Evaluable immunogenicity population. Here, number of participants analyzed signifies participants with valid and determinate hSBA titers for the given strain. Here, N signifies participants with valid and determinate hSBA titers for the given strain at the specified time point. This outcome measure was planned to be analyzed for Group 1 only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 300
Percentage of participants
  PMB3175[A29]:Before Vaccination 1 (N=280) | 31.1 [25.7 to 36.9]
  PMB3175[A29]:1 Month after Vaccination 3 (N=283) | 99.3 [97.5 to 99.9]
  PMB3010[A06]:Before Vaccination 1 (N=275) | 16.0 [11.9 to 20.9]
  PMB3010[A06]:1 Month after Vaccination 3 (N=275) | 92.0 [88.1 to 94.9]
  PMB3040[A07]:Before Vaccination 1 (N=274) | 55.8 [49.7 to 61.8]
  PMB3040[A07]:1 Month after Vaccination 3 (N=277) | 95.7 [92.6 to 97.7]
  PMB824[A12]: Before Vaccination 1 (N=278) | 5.0 [2.8 to 8.3]
  PMB824[A12]:1 Month after Vaccination 3 (N=275) | 71.3 [65.5 to 76.5]
  PMB1672[A15]:Before Vaccination 1 (N=279) | 37.3 [31.6 to 43.2]
  PMB1672[A15]:1 Month after Vaccination 3 (N=279) | 91.8 [87.9 to 94.7]
  PMB1989[A19]:Before Vaccination 1 (N=278) | 28.8 [23.5 to 34.5]
  PMB1989[A19]:1 Month after Vaccination 3 (N=284) | 95.8 [92.7 to 97.8]
  PMB1256[B03]:Before Vaccination 1 (N=277) | 11.2 [7.7 to 15.5]
  PMB1256[B03]:1 Month after Vaccination 3 (N=273) | 86.4 [81.8 to 90.3]
  PMB866[B09]:Before Vaccination 1 (N=277) | 23.5 [18.6 to 28.9]
  PMB866[B09]:1 Month after Vaccination 3 (N=274) | 77.0 [71.6 to 81.9]
  PMB431[B15]:Before Vaccination 1 (N=274) | 43.8 [37.8 to 49.9]
  PMB431[B15]:1 Month after Vaccination 3 (N=276) | 96.7 [93.9 to 98.5]
  PMB648[B16]:Before Vaccination 1 (N=270) | 21.9 [17.1 to 27.3]
  PMB648[B16]:1 Month after Vaccination 3 (N=273) | 78.0 [72.6 to 82.8]

39. Secondary Outcome: Percentage of Participants With hSBA Titers >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, >=1:128 for Each of the 10 Secondary Strains Before First Vaccination and 1 Month After the Third Bivalent rLP2086 Vaccination: Group 1
Time Frame: Before first vaccination, 1 month after third vaccination (Vac)
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 300
Percentage of participants
  Before Vaccination 1: PMB3175[A29] 1:4 (N=280) | 32.9 [27.4 to 38.7]
  1 month after Vac 3: PMB3175[A29] 1:4 (N=283) | 99.3 [97.5 to 99.9]
  Before Vaccination 1: PMB3175[A29] 1:8 (N=280) | 31.1 [25.7 to 36.9]
  1 month after Vac 3: PMB3175[A29] 1:8 (N=283) | 99.3 [97.5 to 99.9]
  Before Vaccination 1: PMB3175[A29] 1:16 (N=280) | 27.9 [22.7 to 33.5]
  1 month after Vac 3: PMB3175[A29] 1:16 (N=283) | 98.9 [96.9 to 99.8]
  Before Vaccination 1: PMB3175[A29] 1:32 (N=280) | 16.1 [12.0 to 20.9]
  1 month after Vac 3: PMB3175[A29] 1:32 (N=283) | 96.8 [94.0 to 98.5]
  Before Vaccination 1: PMB3175[A29] 1:64 (N=280) | 5.7 [3.3 to 9.1]
  1 month after Vac 3: PMB3175[A29] 1:64 (N=283) | 80.9 [75.8 to 85.3]
  Before Vaccination 1: PMB3175[A29] 1:128 (N=280) | 2.1 [0.8 to 4.6]
  1 month after Vac 3: PMB3175[A29] 1:128 (N=283) | 53.0 [47.0 to 58.9]
  Before Vaccination 1: PMB3010[A06] 1:4 (N=275) | 18.9 [14.5 to 24.0]
  1 month after Vac 3: PMB3010[A06] 1:4 (N=275) | 92.4 [88.6 to 95.2]
  Before Vaccination 1: PMB3010[A06] 1:8 (N=275) | 17.5 [13.2 to 22.5]
  1 month after Vac 3: PMB3010[A06] 1:8 (N=275) | 92.4 [88.6 to 95.2]
  Before Vaccination 1: PMB3010[A06] 1:16 (N=275) | 16.0 [11.9 to 20.9]
  1 month after Vac 3: PMB3010[A06] 1:16 (N=275) | 92.0 [88.1 to 94.9]
  Before Vaccination 1: PMB3010[A06] 1:32 (N=275) | 10.5 [7.2 to 14.8]
  1 month after Vac 3: PMB3010 [A06] 1:32 (N=275) | 86.2 [81.5 to 90.0]
  Before Vaccination 1: PMB3010[A06] 1:64 (N=275) | 6.5 [3.9 to 10.1]
  1 month after Vac 3: PMB3010[A06] 1:64 (N=275) | 70.5 [64.8 to 75.9]
  Before Vaccination 1: PMB3010[A06] 1:128 (N=275) | 2.5 [1.0 to 5.2]
  1 month after Vac 3: PMB3010[A06] 1:128 (N=275) | 41.8 [35.9 to 47.9]
  Before Vaccination 1: PMB3040[A07] 1:4 (N=274) | 55.8 [49.7 to 61.8]
  1 month after Vac 3: PMB3040[A07] 1:4 (N=277) | 95.7 [92.6 to 97.7]
  Before Vaccination 1: PMB3040[A07] 1:8 (N=274) | 55.8 [49.7 to 61.8]
  1 month after Vac 3: PMB3040[A07] 1:8 (N=277) | 95.7 [92.6 to 97.7]
  Before Vaccination 1: PMB3040[A07] 1:16 (N=274) | 55.5 [49.4 to 61.5]
  1 month after Vac 3: PMB3040[A07] 1:16 (N=277) | 95.7 [92.6 to 97.7]
  Before Vaccination 1: PMB3040[A07] 1:32 (N=274) | 42.7 [36.8 to 48.8]
  1 month after Vac 3: PMB3040[A07] 1:32 (N=277) | 92.4 [88.6 to 95.2]
  Before Vaccination 1: PMB3040[A07] 1:64 (N=274) | 21.2 [16.5 to 26.5]
  1 month after Vac 3: PMB3040[A07] 1:64 (N=277) | 72.9 [67.3 to 78.1]
  Before Vaccination 1: PMB3040[A07] 1:128 (N=274) | 4.0 [2.0 to 7.1]
  1 month after Vac 3: PMB3040[A07] 1:128 (N=277) | 29.2 [24.0 to 35.0]
  Before Vaccination 1: PMB824[A12] 1:4 (N=278) | 10.4 [7.1 to 14.6]
  1 month after Vac 3: PMB824[A12] 1:4 (N=275) | 73.8 [68.2 to 78.9]
  Before Vaccination 1: PMB824[A12] 1:8 (N=278) | 8.3 [5.3 to 12.2]
  1 month after Vac 3: PMB824[A12] 1:8 (N=275) | 73.5 [67.8 to 78.6]
  Before Vaccination 1: PMB824[A12] 1:16 (N=278) | 5.0 [2.8 to 8.3]
  1 month after Vac 3: PMB824[A12] 1:16 (N=275) | 71.3 [65.5 to 76.5]
  Before Vaccination 1: PMB824[A12] 1:32 (N=278) | 2.2 [0.8 to 4.6]
  1 month after Vac 3: PMB824[A12] 1:32 (N=275) | 46.5 [40.5 to 52.6]
  Before Vaccination 1: PMB824[A12] 1:64 (N=278) | 0.0 [0.0 to 1.3]
  1 month after Vac 3: PMB824[A12] 1:64 (N=275) | 15.6 [11.6 to 20.5]
  Before Vaccination 1: PMB824[A12] 1:128 (N=278) | 0.0 [0.0 to 1.3]
  1 month after Vac 3: PMB824[A12] 1:128 (N=275) | 3.3 [1.5 to 6.1]
  Before Vaccination 1: PMB1672[A15] 1:4 (N=279) | 39.4 [33.7 to 45.4]
  1 month after Vac 3: PMB1672[A15] 1:4 (N=279) | 91.8 [87.9 to 94.7]
  Before Vaccination 1: PMB1672[A15] 1:8 (N=279) | 37.3 [31.6 to 43.2]
  1 month after Vac 3: PMB1672[A15] 1:8 (N=279) | 91.8 [87.9 to 94.7]
  Before Vaccination 1: PMB1672[A15] 1:16 (N=279) | 33.3 [27.8 to 39.2]
  1 month after Vac 3: PMB1672[A15] 1:16 (N=279) | 91.4 [87.5 to 94.4]
  Before Vaccination 1: PMB1672[A15] 1:32 (N=279) | 20.4 [15.9 to 25.6]
  1 month after Vac 3: PMB1672[A15] 1:32 (N=279) | 82.4 [77.5 to 86.7]
  Before Vaccination 1: PMB1672[A15] 1:64 (N=279) | 7.2 [4.4 to 10.9]
  1 month after Vac 3: PMB1672[A15] 1:64 (N=279) | 54.5 [48.4 to 60.4]
  Before Vaccination 1: PMB1672[A15] 1:128 (N=279) | 1.8 [0.6 to 4.1]
  1 month after Vac 3: PMB1672[A15] 1:128 (N=279) | 19.0 [14.6 to 24.1]
  Before Vaccination 1: PMB1989[A19] 1:4 (N=278) | 39.2 [33.4 to 45.2]
  1 month after Vac 3: PMB1989[A19] 1:4 (N=284) | 96.1 [93.2 to 98.1]
  Before Vaccination 1: PMB1989[A19] 1:8 (N=278) | 37.1 [31.4 to 43.0]
  1 month after Vac 3: PMB1989[A19] 1:8 (N=284) | 96.1 [93.2 to 98.1]
  Before Vaccination 1: PMB1989[A19] 1:16 (N=278) | 28.8 [23.5 to 34.5]
  1 month after Vac 3: PMB1989[A19] 1:16 (N=284) | 95.8 [92.7 to 97.8]
  Before Vaccination 1: PMB1989[A19] 1:32 (N=278) | 18.3 [14.0 to 23.4]
  1 month after Vac 3: PMB1989[A19] 1:32 (N=284) | 92.3 [88.5 to 95.1]
  Before Vaccination 1: PMB1989[A19] 1:64 (N=278) | 9.0 [5.9 to 13.0]
  1 month after Vac 3: PMB1989[A19] 1:64 (N=284) | 77.5 [72.2 to 82.2]
  Before Vaccination 1: PMB1989[A19] 1:128 (N=278) | 9.0 [5.9 to 13.0]
  1 month after Vac 3: PMB1989[A19] 1:128 (N=284) | 49.6 [43.7 to 55.6]
  Before Vaccination 1: PMB1256[B03] 1:4 (N=277) | 13.0 [9.3 to 17.5]
  1 month after Vac 3: PMB1256[B03] 1:4 (N=273) | 86.8 [82.2 to 90.6]
  Before Vaccination 1: PMB1256[B03] 1:8 (N=277) | 11.2 [7.7 to 15.5]
  1 month after Vac 3: PMB1256[B03] 1:8 (N=273) | 86.4 [81.8 to 90.3]
  Before Vaccination 1: PMB1256[B03] 1:16 (N=277) | 10.1 [6.8 to 14.3]
  1 month after Vac 3: PMB1256[B03] 1:16 (N=273) | 85.3 [80.6 to 89.3]
  Before Vaccination 1: PMB1256[B03] 1:32 (N=277) | 7.6 [4.8 to 11.4]
  1 month after Vac 3: PMB1256[B03] 1:32 (N=273) | 78.4 [73.0 to 83.1]
  Before Vaccination 1: PMB1256[B03] 1:64 (N=277) | 4.7 [2.5 to 7.9]
  1 month after Vac 3: PMB1256[B03] 1:64 (N=273) | 56.4 [50.3 to 62.4]
  Before Vaccination 1: PMB1256[B03] 1:128 (N=277) | 1.1 [0.2 to 3.1]
  1 month after Vac 3: PMB1256[B03] 1:128 (N=273) | 30.8 [25.3 to 36.6]
  Before Vaccination 1: PMB866[B09] 1:4 (N=277) | 24.5 [19.6 to 30.1]
  1 month after Vac 3: PMB866[B09] 1:4 (N=274) | 78.5 [73.1 to 83.2]
  Before Vaccination 1: PMB866[B09] 1:8 (N=277) | 23.5 [18.6 to 28.9]
  1 month after Vac 3: PMB866[B09] 1:8 (N=274) | 77.0 [71.6 to 81.9]
  Before Vaccination 1: PMB866[B09] 1:16 (N=277) | 18.8 [14.3 to 23.9]
  1 month after Vac 3: PMB866[B09] 1:16 (N=274) | 73.4 [67.7 to 78.5]
  Before Vaccination 1: PMB866[B09] 1:32 (N=277) | 11.9 [8.3 to 16.3]
  1 month after Vac 3: PMB866[B09] 1:32 (N=274) | 52.6 [46.5 to 58.6]
  Before Vaccination 1: PMB866[B09] 1:64 (N=277) | 4.7 [2.5 to 7.9]
  1 month after Vac 3: PMB866[B09] 1:64 (N=274) | 27.7 [22.5 to 33.4]
  Before Vaccination 1: PMB866[B09] 1:128 (N=277) | 1.1 [0.2 to 3.1]
  1 month after Vac 3: PMB866[B09] 1:128 (N=274) | 12.8 [9.1 to 17.3]
  Before Vaccination 1: PMB431[B15] 1:4 (N=274) | 44.9 [38.9 to 51.0]
  1 month after Vac 3: PMB431[B15] 1:4 (N=276) | 97.1 [94.4 to 98.7]
  Before Vaccination 1: PMB431[B15] 1:8 (N=274) | 43.8 [37.8 to 49.9]
  1 month after Vac 3: PMB431[B15] 1:8 (N=276) | 96.7 [93.9 to 98.5]
  Before Vaccination 1: PMB431[B15] 1:16 (N=274) | 41.2 [35.4 to 47.3]
  1 month after Vac 3: PMB431[B15] 1:16 (N=276) | 96.7 [93.9 to 98.5]
  Before Vaccination 1: PMB431[B15] 1:32 (N=274) | 23.7 [18.8 to 29.2]
  1 month after Vac 3: PMB431[B15] 1:32 (N=276) | 84.4 [79.6 to 88.5]
  Before Vaccination 1: PMB431[B15] 1:64 (N=274) | 8.0 [5.1 to 11.9]
  1 month after Vac 3: PMB431[B15] 1:64 (N=276) | 56.5 [50.4 to 62.5]
  Before Vaccination 1: PMB431[B15] 1:128 (N=274) | 1.5 [0.4 to 3.7]
  1 month after Vac 3: PMB431[B15] 1:128 (N=276) | 22.5 [17.7 to 27.9]
  Before Vaccination 1: PMB648[B16] 1:4 (N=270) | 24.4 [19.4 to 30.0]
  1 month after Vac 3: PMB648[B16] 1:4 (N=273) | 79.1 [73.8 to 83.8]
  Before Vaccination 1: PMB648[B16] 1:8 (N=270) | 21.9 [17.1 to 27.3]
  1 month after Vac 3: PMB648[B16] 1:8 (N=273) | 78.0 [72.6 to 82.8]
  Before Vaccination 1: PMB648[B16] 1:16 (N=270) | 18.9 [14.4 to 24.1]
  1 month after Vac 3: PMB648[B16] 1:16 (N=273) | 76.6 [71.1 to 81.5]
  Before Vaccination 1: PMB648[B16] 1:32 (N=270) | 11.9 [8.2 to 16.3]
  1 month after Vac 3: PMB648[B16] 1:32 (N=273) | 61.2 [55.1 to 67.0]
  Before Vaccination 1: PMB648[B16] 1:64 (N=270) | 7.4 [4.6 to 11.2]
  1 month after Vac 3: PMB648[B16] 1:64 (N=273) | 34.4 [28.8 to 40.4]
  Before Vaccination 1: PMB648[B16] 1:128 (N=270) | 1.9 [0.6 to 4.3]
  1 month after Vac 3: PMB648[B16] 1:128 (N=273) | 16.8 [12.6 to 21.8]

40. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) for Each of the 10 Secondary Strains Before First Vaccination and 1 Month After the Third Bivalent rLP2086 Vaccination: Group 1
Time Frame: Before first vaccination, 1 month after third vaccination
Population: Evaluable immunogenicity population. Here, number of participants analyzed signifies participants with valid and determinate hSBA titers for the given strain. Here, N signifies participants with valid and determinate assay results for the given antigen or strain. This outcome measure was planned to be analyzed for Group 1 only.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 300
Titers
  PMB3175[A29]:Before Vaccination 1 (N=280) | 7.1 [6.4 to 8.0]
  PMB3175[A29]:1 Month after Vaccination 3 (N=283) | 96.3 [86.9 to 106.9]
  PMB3010[A06]:Before Vaccination 1 (N=275) | 10.3 [9.5 to 11.2]
  PMB3010[A06]:1 Month after Vaccination 3 (N=275) | 69.9 [61.8 to 79.1]
  PMB3040[A07]:Before Vaccination 1 (N=274) | 13.9 [12.0 to 16.0]
  PMB3040[A07]:1 Month after Vaccination 3 (N=277) | 60.4 [54.6 to 66.8]
  PMB824[A12]: Before Vaccination 1 (N=278) | 8.4 [8.2 to 8.6]
  PMB824[A12]:1 Month after Vaccination 3 (N=275) | 20.6 [18.8 to 22.6]
  PMB1672[A15]:Before Vaccination 1 (N=279) | 8.0 [7.1 to 9.0]
  PMB1672[A15]:1 Month after Vaccination 3 (N=279) | 43.1 [38.4 to 48.4]
  PMB1989[A19]:Before Vaccination 1 (N=278) | 12.1 [11.1 to 13.3]
  PMB1989[A19]:1 Month after Vaccination 3 (N=284) | 87.3 [77.7 to 98.0]
  PMB1256[B03]:Before Vaccination 1 (N=277) | 5.1 [4.7 to 5.6]
  PMB1256[B03]:1 Month after Vaccination 3 (N=273) | 49.8 [42.2 to 58.7]
  PMB866[B09]:Before Vaccination 1 (N=277) | 6.1 [5.5 to 6.7]
  PMB866[B09]:1 Month after Vaccination 3 (N=274) | 23.3 [19.9 to 27.1]
  PMB431[B15]:Before Vaccination 1 (N=274) | 9.1 [8.1 to 10.3]
  PMB431[B15]:1 Month after Vaccination 3 (N=276) | 49.4 [44.6 to 54.8]
  PMB648[B16]:Before Vaccination 1 (N=270) | 6.2 [5.5 to 6.9]
  PMB648[B16]:1 Month after Vaccination 3 (N=273) | 26.5 [22.8 to 30.8]

41. Secondary Outcome: Percentage of Participants Achieving Composite hSBA Titer >=Lower Limit of Quantitation for All 4 Primary Strains Before First Vaccination and 1 Month After Second Bivalent rLP2086 Vaccination: Group 1
Time Frame: Before vaccination 1, 1 Month after Vaccination 2
Population: Evaluable immunogenicity population. Here, N signifies participants valid and determinate hSBA results on all 4 strains at the given time point. This outcome measure was planned to be analyzed for Group 1 only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 1723
Percentage of participants
  Before First Vaccination (N=1612) | 7.3 [6.0 to 8.6]
  1 Month after Vaccination 2 (N=1620) | 64.5 [62.1 to 66.8]

42. Secondary Outcome: Percentage of Participants Achieving at Least a 4-Fold Increase in hSBA Titer for Each of the 4 Primary Strains Before First Vaccination to 1 Month After the Second Bivalent rLP2086 Vaccination: Group 1
Time Frame: One month after second Bivalent rLP2086 vaccination
Population: Evaluable immunogenicity population. Here, N signifies participants with valid and determinate hSBA titers for the given strain at both the specified time point. This outcome measure was planned to be analyzed for Group 1 only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 1723
Percentage of participants
  PMB80[A22] (N=1679) | 66.9 [64.6 to 69.2]
  PMB2001[A56] (N=1637) | 85.9 [84.1 to 87.5]
  PMB2948[B24] (N=1658) | 67.9 [65.6 to 70.2]
  PMB2707[B44] (N=1686) | 55.5 [53.1 to 57.9]

43. Secondary Outcome: Percentage of Participants With hSBA Titers >=LLOQ for 4 Primary Test Strains Before First Vaccination, 1 Month After Second and Third Bivalent rLP2086 Vaccination: Group 1
Time Frame: Before Vaccination (Vac) 1, 1 Month after Vac 2, 3
Population: Evaluable immunogenicity population. Here, N signifies participants with valid and determinate hSBA titers for the given strain at the specified time point. This outcome measure was planned to be analyzed for Group 1 only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 1723
Percentage of participants
  Before Vac 1: PMB80[A22] 1:16 (N=1704) | 33.6 [31.3 to 35.9]
  1 month after Vac 2: PMB80[A22] 1:16 (N=1697) | 84.7 [82.9 to 86.4]
  1 month after Vac 3: PMB80[A22] 1:16 (N=1714) | 93.5 [92.2 to 94.6]
  Before Vac 1: PMB2001[A56] 1:8 (N=1657) | 32.2 [29.9 to 34.5]
  1 month after Vac 2: PMB2001[A56] 1:8) (N=1701) | 97.4 [96.5 to 98.1]
  1 month after Vac 3: PMB2001[A56] 1:8 (N=1708) | 99.4 [98.9 to 99.7]
  Before Vac 1: PMB2948[B24] 1:8 (N=1696) | 33.1 [30.9 to 35.4]
  1 month after Vac 2: PMB2948[B24] 1:8 (N=1685) | 86.5 [84.7 to 88.1]
  1 month after Vac 3:PMB2948[B24] 1:8 (N=1702) | 95.1 [93.9 to 96.0]
  Before Vac 1: PMB2707[B44] 1:8 (N=1716) | 11.0 [9.6 to 12.6]
  1 month after Vac 2: PMB2707[B44] 1:8 (N=1693) | 68.3 [66.1 to 70.6]
  1 month after Vac 3: PMB2707[B44] 1:8 (N=1703) | 87.4 [85.8 to 89.0]

44. Secondary Outcome: Percentage of Participants With hSBA Titers >=1:4,>=1:8,>=1:16,>=1:32,>=1:64,>=1:128 for 4 Primary Test Strains Before First Vaccination, 1 Month After Second and Third Bivalent rLP2086 Vaccination: Group 1
Description: Results for PMB80[A22] 1:16, PMB2001[A56] 1:8, PMB2948[B24] 1:8 and PMB2707[B44] 1:8 are reported under secondary endpoint 'Percentage of Participants With hSBA Titers >=LLOQ for 4 Primary Test Strains Before First Vaccination, 1 Month After Second and Third Bivalent rLP2086 Vaccination: Group 1'.
Time Frame: Before Vaccination (Vac) 1, 1 Month after Vac 2, 3
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 1723
Percentage of participants
  Before Vac 1: PMB80[A22] 1:4 (N=1704) | 42.1 [39.7 to 44.5]
  1 month after Vac 2: PMB80[A22] 1:4 (N=1697) | 86.2 [84.5 to 87.8]
  1 month after Vac 3: PMB80[A22] 1:4 (N=1714) | 94.3 [93.1 to 95.3]
  Before Vac 1: PMB80[A22] 1:8 (N=1704) | 38.8 [36.5 to 41.2]
  1 month after Vac 2: PMB80[A22] 1:8 (N=1697) | 85.7 [83.9 to 87.3]
  1 month after Vac 3: PMB80[A22] 1:8 (N=1714) | 94.1 [92.9 to 95.2]
  Before Vac 1: PMB80[A22] 1:32 (N=1704) | 19.7 [17.8 to 21.6]
  1 month after Vac 2: PMB80[A22] 1:32 (N=1697) | 71.2 [69.0 to 73.3]
  1 month after Vac 3: PMB80[A22] 1:32 (N=1714) | 85.5 [83.8 to 87.2]
  Before Vac 1: PMB80[A22] 1:64 (N=1704) | 9.6 [8.3 to 11.1]
  1 month after Vac 2: PMB80[A22] 1:64 (N=1697) | 49.9 [47.4 to 52.3]
  1 month after Vac 3: PMB80[A22] 1:64 (N=1714) | 64.4 [62.1 to 66.7]
  Before Vac 1: PMB80[A22] 1:128 (N=1704) | 3.4 [2.6 to 4.4]
  1 month after Vac 2: PMB80[A22] 1:128 (N=1697) | 29.9 [27.8 to 32.2]
  1 month after Vac 3: PMB80[A22] 1:128 (N=1714) | 41.7 [39.4 to 44.1]
  Before Vac 1: PMB2001[A56] 1:4 (N=1657) | 35.9 [33.6 to 38.3]
  1 month after Vac 2: PMB2001[A56] 1:4 (N=1701) | 97.8 [97.0 to 98.5]
  1 month after Vac 3: PMB2001[A56] 1:4 (N=1708) | 99.4 [98.9 to 99.7]
  Before Vac 1: PMB2001[A56] 1:16 (N=1657) | 30.4 [28.2 to 32.7]
  1 month after Vac 2: PMB2001[A56] 1:16 (N=1701) | 97.1 [96.1 to 97.8]
  1 month after Vac 3: PMB2001[A56] 1:16 (N=1708) | 99.2 [98.7 to 99.6]
  Before Vac 1: PMB2001[A56] ] 1:32 (N=1657) | 24.4 [22.3 to 26.5]
  1 month after Vac 2: PMB2001[A56] 1:32 (N=1701) | 92.8 [91.4 to 94.0]
  1 month after Vac 3: PMB2001[A56] 1:32 (N=1708) | 97.2 [96.4 to 98.0]
  Before Vac 1: PMB2001[A56] 1:64 (N=1657) | 16.4 [14.6 to 18.2]
  1 month after Vac 2 :PMB2001[A56] 1:64 (N=1701) | 80.8 [78.9 to 82.7]
  1 month after Vac 3 :PMB2001[A56] 1:64 (N=1708) | 90.5 [89.0 to 91.9]
  Before Vac 1: PMB2001[A56] 1:128 (N=1657) | 7.1 [5.9 to 8.5]
  1 month after Vac 2: PMB2001[A56] 1:128 (N=1701) | 56.6 [54.2 to 58.9]
  1 month after Vac 3: PMB2001[A56] 1:128 (N=1708) | 73.7 [71.5 to 75.7]
  Before Vac 1: PMB2948[B24] 1:4 (N=1696) | 35.0 [32.7 to 37.3]
  1 month after Vac 2: PMB2948[B24] 1:4 (N=1685) | 87.2 [85.5 to 88.7]
  1 month after Vac 3: PMB2948[B24] 1:4 (N=1702) | 95.8 [94.8 to 96.7]
  Before Vac 1: PMB2948[B24] 1:16 (N=1696) | 29.5 [27.3 to 31.7]
  1 month after Vac 2: PMB2948[B24] 1:16 (N=1685) | 83.7 [81.9 to 85.5]
  1 month after Vac 3: PMB2948[B24] 1:16 (N=1702) | 93.2 [91.9 to 94.3]
  Before Vac 1: PMB2948[B24] 1:32 (N=1696) | 18.1 [16.3 to 20.0]
  1 month after Vac 2: PMB2948[B24] 1:32 (N=1685) | 65.6 [63.3 to 67.8]
  1 month after Vac 3: PMB2948[B24] 1:32 (N=1702) | 75.1 [73.0 to 77.2]
  Before Vac 1: PMB2948[B24] 1:64 (N=1696) | 8.4 [7.1 to 9.8]
  1 month after Vac 2: PMB2948[B24] 1:64 (N=1685) | 40.4 [38.0 to 42.7]
  1 month after Vac 3: PMB2948[B24] 1:64 (N=1702) | 48.8 [46.4 to 51.2]
  Before Vac 1: PMB2948[B24] 1:128 (N=1696) | 3.3 [2.5 to 4.3]
  1 month after Vac 2: PMB2948[B24] 1:128 (N=1685) | 22.8 [20.9 to 24.9]
  1 month after Vac 3: PMB2948[B24] 1:128 (N=1702) | 27.8 [25.7 to 30.0]
  Before Vac 1: PMB2707[B44] 1:4 (N=1716) | 14.5 [12.8 to 16.2]
  1 month after Vac 2: PMB2707[B44] 1:4 (N=1693) | 71.5 [69.3 to 73.7]
  1 month after Vac 3: PMB2707[B44] 1:4 (N=1703) | 89.7 [88.1 to 91.1]
  Before Vac 1: PMB2707[B44] 1:16 (N=1716) | 7.8 [6.5 to 9.1]
  1 month after Vac 2: PMB2707[B44] 1:16 (N=1693) | 61.0 [58.6 to 63.3]
  1 month after Vac 3: PMB2707[B44] 1:16 (N=1703) | 83.3 [81.4 to 85.0]
  Before Vac 1: PMB2707[B44] 1:32 (N=1716) | 4.3 [3.4 to 5.4]
  1 month after Vac 2: PMB2707[B44] 1:32 (N=1693) | 41.9 [39.6 to 44.3]
  1 month after Vac 3: PMB2707[B44] 1:32 (N=1703) | 67.1 [64.8 to 69.3]
  Before Vac 1: PMB2707[B44] 1:64 (N=1716) | 2.3 [1.6 to 3.1]
  1 month after Vac 2: PMB2707[B44] 1:64 (N=1693) | 30.3 [28.1 to 32.6]
  1 month after Vac 3: PMB2707[B44] 1:64 (N=1703) | 49.8 [47.4 to 52.2]
  Before Vac 1: PMB2707[B44] 1:128 (N=1716) | 0.8 [0.4 to 1.3]
  1 month after Vac 2: PMB2707[B44] 1:128 (N=1693) | 21.0 [19.1 to 23.0]
  1 month after Vac 3: PMB2707[B44] 1:128 (N=1703) | 32.1 [29.9 to 34.4]

45. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) for 4 Primary Test Strains Before First Vaccination, 1 Month After Second and Third Bivalent rLP2086 Vaccination: Group 1
Time Frame: Before Vaccination (Vac) 1, 1 Month after Vac 2, 3
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 1723
Titer
  PMB80[A22]: Before Vac 1 (N=1704) | 12.8 [12.3 to 13.3]
  PMB80[A22]: 1 Month after Vac 2 (N=1697) | 49.0 [46.2 to 52.1]
  PMB80[A22]: 1 Month after Vac 3 (N=1714) | 74.3 [70.2 to 78.6]
  PMB2001[A56]: Before Vac 1 (N=1657) | 8.8 [8.3 to 9.3]
  PMB2001[A56]: 1 Month after Vac 2 (N=1701) | 114.3 [107.9 to 121.0]
  PMB2001[A56]: 1 Month after Vac 3 (N=1708) | 176.7 [167.8 to 186.1]
  PMB2948[B24]: Before Vac 1 (N=1696) | 7.6 [7.3 to 8.0]
  PMB2948[B24]: 1 Month after Vac 2 (N=1685) | 35.8 [33.7 to 38.2]
  PMB2948[B24]: 1 Month after Vac 3 (N=1702) | 49.5 [46.8 to 52.4]
  PMB2707[B44]: Before Vac 1 (N=1716) | 4.8 [4.7 to 4.9]
  PMB2707[B44]: 1 Month after Vac 2 (N=1693) | 22.6 [20.9 to 24.4]
  PMB2707[B44]: 1 Month after Vac 3 (N=1703) | 47.6 [44.2 to 51.3]

46. Secondary Outcome: Percentage of Participants Achieving at Least a 3-Fold Increase in hSBA Titer for 4 Primary Test Strains Before First Vaccination to 1 Month After Third Bivalent rLP2086 Vaccination
Time Frame: One month after third bivalent rLP2086 vaccination
Population: Data was not reported because 3-fold rise analyses was not performed as per change in planned analysis.
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 0

47. Secondary Outcome: Percentage of Participants Achieving at Least a 2-Fold Increase in hSBA Titer for 4 Primary Test Strains Before First Vaccination to 1 Month After the Third Bivalent rLP2086 Vaccination: Group 1
Time Frame: One month after third bivalent rLP2086 vaccination
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 rLP2086
Number analyzed (Participants) | 1723
Percentage of participants
  PMB80[A22]: 1 Month after Vac 3 (N=1695) | 89.0 [87.4 to 90.4]
  PMB2001[A56]: 1 Month after Vac 3 (N=1642) | 95.3 [94.2 to 96.3]
  PMB2948[B24]: 1 Month after Vac 3 (N=1675) | 87.1 [85.4 to 88.7]
  PMB2707[B44]: 1 Month after Vac 3(N=1696) | 81.8 [79.9 to 83.6]

ADVERSE EVENTS:
Time Frame: AEs/SAEs: recorded from first vaccination through 6 months after third vaccination. Participants recorded pre-specified reactogenicity events (local reactions, systemic events) in electronic diary within 7 days after first, second and third vaccination
Description: All AEs collected on case report form are shown below as having been collected via non-systematic assessment. All events reported via electronic diary (reactogenicity events) are shown below as having been collected via systematic assessment. Reactogenicity events are grouped by all severities and doses combined.
Arm/Group | Group 1 rLP2086 | Group 2 Saline
Serious Adverse Events (participants affected / at risk) | 33/2471 | 11/822
Other Adverse Events (participants affected / at risk) | 2193/2471 | 567/822
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 rLP2086 (N=2471) | Group 2 Saline (N=822)
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 1
Cystitis (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Otosalpingitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 2
Benign intracranial hypertension (Nervous system disorders) | 1 | 0
Dystonia (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 4 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Dissociative disorder (Psychiatric disorders) | 1 | 0
Eating disorder (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Group 1 rLP2086 (N=2471) | Group 2 Saline (N=822)
Injection site pain (General disorders) | 46 | 6
Fatigue (General disorders) | 12 | 10
Upper respiratory tract infection (Infections and infestations) | 98 | 29
Nasopharyngitis (Infections and infestations) | 77 | 33
Urinary tract infection (Infections and infestations) | 45 | 10
Pharyngitis (Infections and infestations) | 37 | 10
Gastroenteritis (Infections and infestations) | 33 | 12
Tonsillitis (Infections and infestations) | 19 | 11
Bronchitis (Infections and infestations) | 12 | 10
Fall (Injury, poisoning and procedural complications) | 31 | 6
Ligament sprain (Injury, poisoning and procedural complications) | 22 | 11
Headache (Nervous system disorders) | 55 | 10
Pain at injection site - Any (reactogenicity event) (Skin and subcutaneous tissue disorders) | 2184/2438 | 147/808
Redness -Any (reactogenicity event) (Skin and subcutaneous tissue disorders) | 537/2438 | 8/808
Swelling -Any (reactogenicity event) (Skin and subcutaneous tissue disorders) | 612/2438 | 8/808
Fever >=38.0 degrees C -Any (reactogenicity event) (General disorders) | 108/2432 | 14/807
Vomiting - Any (reactogenicity event) (General disorders) | 130/2438 | 37/808
Diarrhea-Any (reactogenicity event) (General disorders) | 497/2438 | 158/808
Headache - Any (reactogenicity event) (General disorders) | 1440/2438 | 391/808
Fatigue -Any (reactogenicity event) (General disorders) | 1576/2438 | 411/808
Chills - Any (reactogenicity event) (General disorders) | 697/2438 | 133/808
Muscle pain -Any (reactogenicity event) (General disorders) | 916/2438 | 170/808
Joint pain -Any (reactogenicity event) (General disorders) | 723/2438 | 136/808

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.